CLINICAL TRIAL: NCT02618291
Title: Efficacy of a an Active Geriatric Evaluation (AGE Tool) for Geriatric Syndromes to Prevent Functional Decline in Elderly Patients in Family Medicine: a Pragmatic Cluster Randomized Trial
Brief Title: Efficacy of an Active Geriatric Evaluation for Geriatric Syndromes to Prevent Functional Decline in Family Medicine
Acronym: AGE3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Nicolas Senn, Head of research and de development centre, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 32003B_159863/1
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Geriatric Syndrome; Functional Ability
Keywords: primary health care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Geriatric Evaluation (AGE tool) (Experimental): The Active Geriatric Evaluation is a comprehensive assessment and management tool consisting of a 20-minute clinical screening instrument (Brief Assessment Tool, BAT) to identify 8 geriatric syndromes, and complementary diagnostic evaluations and propositions of management & treatment for each syndrome.
  Interventions: Other: Active Geriatric Evaluation (AGE tool)
- Usual care (Active Comparator): No specific intervention will be provided to the patients, except what family practitioners (FPs) usually do. In this regard, it is possible that some FPs might use structured interventions similar to the AGE tool. This will be neither encouraged nor discouraged. FPs in the "usual care" arm will be asked to perform one BAT after 2 years of follow-up, at the final patient visit.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Active Geriatric Evaluation (AGE tool) — Yearly administration of the brief assessment tool (BAT). Once the presence of one or more geriatric syndromes is suspected using the brief assessment tool, a management strategy is proposed. It is divided in two distinct steps: 1) perform additional tests to confirm or exclude the diagnosis and 2) to propose specific management attitudes. All proposed attitudes are based on literature review and geriatrician expertise. The FP remains free to follow the proposed attitudes.
  Other Names: Active geriatric evaluation
  Arms: Active Geriatric Evaluation (AGE tool)
Other: Usual care — No specific intervention will be provided to the patients, except what family practitioners (FPs) usually do. In this regard, it is possible that some FPs might use structured interventions similar to the AGE tool. This will be neither encouraged nor discouraged. FPs in the "usual care" arm will be asked to perform one BAT after 2 years of follow-up, at the final patient visit.
  Arms: Usual care

SUMMARY:
This study aims to test the efficacy of a comprehensive assessment and management tool (AGE: Active Geriatric Evaluation) for geriatric syndromes to prevent functional decline in elderly patients followed in family medicine. Family practitioners will be randomised either to the intervention, consisting of a yearly screening for eight geriatric syndromes accompanied by a management plan in case of positive screening, or to usual care. Level of functioning and quality of life of patients in both arms will be assessed over two years.

DETAILED DESCRIPTION:
The ageing of the population is associated to a rapid increase of chronic conditions and more specifically geriatric syndromes for which the health care system is largely unprepared. Being in frontline of this huge arising burden, family practitioners (FP) will need adapted tools to identify and manage elderly patients with complex needs and prevent functional decline while improving quality of life. It is however well recognized that effective and efficient evidence-based interventions adapted to the primary care setting are lacking. The AGE program (Active Geriatric Evaluation) was launched in 2011 and aimed at developing a comprehensive assessment and management tool for FP's to better identify and manage geriatric syndromes. The AGE tool consists of a 20-minute clinical screening instrument (Brief Assessment Tool, BAT), which performances for identifying geriatric syndromes was already assessed in general practice along the AGE program, and a comprehensive approach that encompasses: complementary diagnostic evaluations and propositions of management & treatment for each syndrome. The efficacy and efficiency of the AGE tool for preventing functional decline was never assessed in real life settings of general practice.

The aim of the study is to determine whether a comprehensive tool combining a brief assessment tool (BAT) for the early diagnosis of geriatric syndromes with a structured diagnostic and management strategy impacts on the functional decline and quality of life of elderly patients.

Design: Two-arm open label cluster randomized trial in FP practices, randomization unit: FP

Participants and setting: FP's and their patients aged ≥ 75 years in the French part of Switzerland. In total: 40 FP's (2x20) and 400 patients (2 x 200)

Intervention: Active Geriatric Evaluation. Controls: Usual care provided by FP's. Duration of study: 3 years (2 years of follow-up). Expected outcomes:functional ability of patients in the intervention arm ,measured through the activities of daily living, will be conserved compared to patients in the usual care arm.

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 years or more
* Consider the enrolling physician as his/her reference FP
* Able to understand French
* Living at home (not in institutions)
* Visited his/her FP at least twice during the past year
* Giving signed informed consent (or, in the absence of discerning capacity, giving assent in the presence of a surrogate signing the consent form)

Exclusion Criteria:

* Having had a geriatric or specialized memory consultation in the past 3 months (including assessment during rehabilitation)
* Planning to leave the study area or to change of FP in the next 2 years

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 429 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Instrumental Activities of Daily Living (IADL) | 2 years
  Proportion of patients losing at least 1 instrumental IADL (8 items developed to assess functional status)
Basic Activities of Daily Living (ADL) | 2 years
  Proportion of patients losing at least 1 basic ADL (6 items developed to assess functional status)

SECONDARY OUTCOMES:
Incidence of hospital admissions | During 2 years
  Number of hospital admissions per patient per year
Incidence of institutionalization | During 2 years
  Number of institutionalization per patient per year
Incidence of emergency visits | During 2 years
  Number of emergency visits per patient per year
Incidence of outpatient visits | During 2 years
  Number of outpatient visits to GP per patient per year
Health related quality of life (WHOQOL-OLD) score | 2 years
  questionnaire composed of 24 items. This broadly validated instrument is composed of six facets: 1) Sensory abilities, 2) Autonomy, 3) Past, present and future activities, 4) Social participation, 5) Death and dying and 6) Intimacy

OTHER OUTCOMES:
Adhesion to Active Geriatric Evaluation Tool | 2 years
  Proportion of GPs completing the difference sections of the Active Geriatric Evaluation Tool
Total cost | 2 years
  Comparison, by arm, of total cost, corresponding to the sum of costs billed by FPs, drug prescriptions, hospital and institutional admission costs

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Senn, MD PhD, Principal Investigator — Department of community medicine and ambulatory care, University of Lausanne
Locations (1):
- Department of Ambulatory Care and Community Medicine, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Mueller Y, Schwarz J, Monod S, Locatelli I, Senn N. Use of standardized brief geriatric evaluation compared with routine care in general practice for preventing functional decline: a pragmatic cluster-randomized trial. CMAJ. 2021 Aug 23;193(33):E1289-E1299. doi: 10.1503/cmaj.202887. PMID 34426445
- [Derived] Schnegg D, Senn N, Bugnon O, Schwarz J, Mueller Y. Drug Prescription in Older Swiss Men and Women Followed in Family Medicine. Drugs Real World Outcomes. 2020 Mar;7(1):87-95. doi: 10.1007/s40801-019-00175-6. PMID 31845213

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT02618291/SAP_000.pdf
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02618291/Prot_001.pdf